CLINICAL TRIAL: NCT04550598
Title: Effects of High-definition Transcranial Electrical Stimulation in Patients With Fibromyalgia
Brief Title: High-definition Transcranial Electrical Stimulation for Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Ministry of Health and Welfare (Ambiguous)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202004140
Record Dates: First submitted 2020-08-20; First posted 2020-09-16 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Transcranial electrical stimulation; Analgesic effect
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HD-tCES (Experimental): The experiment group will receive active HD-tCES.
  Interventions: Device: HD-tCES
- Sham HD-tCES (Sham Comparator): The sham control group will receive sham HD-tCES.
  Interventions: Device: Sham HD-tCES

INTERVENTIONS:
Device: HD-tCES — The high definition transcranial electrical stimulation was applied using a 1*4 ring electrode configuration. The electrode will be applied at the left M1 or contralateral to pain side. The anodal electrode was placed on the C3/C4, and the remaining 4 cathodal electrodes were placed in a radius of approximately 7.5 cm from anode (Cz, F3, T7, and P3 on the left hemisphere or Cz, F4, T8, and P4 on the right hemisphere). HD-tCES will be applied for 20 minutes at an intensity of 1.0 mA direct current stimulation and a specific-added waveform each time, 5 times a week, lasting for 2 weeks.
  Arms: HD-tCES
Device: Sham HD-tCES — The high definition transcranial electrical stimulation was applied using a 1*4 ring electrode configuration. The electrode will be applied at the left M1 or contralateral to pain side. The anodal electrode was placed on the C3/C4, and the remaining 4 cathodal electrodes were placed in a radius of approximately 7.5 cm from anode (Cz, F3, T7, and P3 on the left hemisphere or Cz, F4, T8, and P4 on the right hemisphere). Sham HD-tCES will consist of a 5-second ramp up to 1.0 mA direct current stimulation and a specific-added waveform followed immediately by a 5-second ramp down, no current in the middle 19 minutes 40 seconds, and a ramp-up and ramp-down period during the last 10 seconds.
  Arms: Sham HD-tCES

SUMMARY:
Transcranial electrical stimulation (tCES) is a non-invasive and safe treatment, which uses a low direct current or alternating current to change the excitability of the cerebral cortex. The tCES has been applied in clinical trials related to rehabilitation research in recent years, and the safety and effectiveness have also been established. However, the existing tCES products effect on the whole brain networks and lack special waveforms. The investigators developed a wearable high-definition tCES (HD-tCES) with special waveforms. This novel stimulation system will result in more precise and focal stimulation of selected brain regions with special waveforms to display better neuromodulation performance. In this study, the investigators will preliminarily examine the effects and safety of the HD-tCES in patients with fibromyalgia. The investigators expect that the HD-tCES will relief pain, improve sleep quality, emotion, and general health of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. With a diagnosis of fibromyalgia.
2. Age ≥ 20 years.
3. A mean pain score ≥ 4 on a 11-point numeric rating scale during the 2 weeks preceding the trial.

Exclusion Criteria:

1. Intolerance to electrical stimulation.
2. A history of arrhythmia.
3. Implantable medical electronic devices (e.g., like pacemaker).
4. Metal implants in the head or neck.
5. Wounds on the skin of head.
6. A history of brain surgery or severe brain trauma.
7. Severe cognitive or psychiatric disorders (e.g., schizophrenia, depression or bipolar disorder).
8. A history of seizure or other brain pathology.
9. Drug or alcohol abuse.
10. Malignant neoplasm or rheumatism disorder (e.g., SLE, RA, AS, IBD)
11. Pregnancy.
12. Change in medication of fibromyalgia within 1 week prior the trial.
13. Pregnant or breastfeeding women.
14. Intra-cerebral lesions (such as brain tumors, arteriovenous tumors).
15. History of encephalitis or meningitis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Numerical Rating Scale (NRS) after intervention | Baseline (within 7 days ahead to the 1st intervention session), each intervention session in 2 weeks, and after 2-week intervention (within 7 days after the last intervention session)
  The NRS is the simplest and most commonly used numeric scale in which the patient rates the pain from 0 (no pain) to 10 (worst pain).
Change from baseline in the Impact Questionnaire (FIQ) after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 2-week intervention (within 7 days after the last intervention session)
  The FIQ is a brief 10-item, self-administered instrument that measures physical functioning, work status, depression, anxiety, sleep, pain, stiffness, fatigue, and well being.

SECONDARY OUTCOMES:
Change from baseline pressure pain threshold after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 2-week intervention (within 7 days after the last intervention session)
  The pressure pain threshold is defined as the minimum force applied which induces pain. The pressure pain threshold of bilateral trapeziuses, lateral epicondyle of humeri, greater trochanters, and knees will be measured.
Change from baseline in the Beck Depression Inventory Second Edition (BDI-II) after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 2-week intervention (within 7 days after the last intervention session)
  The BDI-II is a 21-item self-report questionnaire that measures major depression symptoms according to diagnostic criteria listed in the Diagnostic and Statistical Manual for Mental Disorders.
Change from baseline in the Beck Anxiety Inventory (BAI) after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 2-week intervention (within 7 days after the last intervention session)
  The BAI is a 21-question multiple-choice self-report inventory that measures the severity of anxiety.
Change from baseline in the Pittsburgh Sleep Quality Index (PSQI) after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 2-week intervention (within 7 days after the last intervention session)
  The PSQI is a 19-item self-report questionnaire that assesses sleep quality.
Change from baseline Tau protein & beta amyloid protein after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 2-week intervention (within 7 days after the last intervention session)
  Tau protein and beta amyloid protein can be the biomarkers of the patient's sleep quality.
Incidence of treatment-emergent adverse events | Within 10 minutes after each intervention session (a total of 10 sessions, 5 sessions/week, lasting 2 weeks)
  Immediately after each HD-tCES stimulation, the patient will be questioned about eventual side effect.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan